CLINICAL TRIAL: NCT04896294
Title: The Effect of Toothpastes Containing Ca-hydroxyapatite, Fluoroapatite, and Mg-Zn-hydroxyapatite on Dentin Hypersensitivity: a Randomized Clinical Trial
Brief Title: Ca-hydroxyapatite, Fluoroapatite, and Mg-Zn-hydroxyapatite for Dentin Hypersensitivity Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18081210
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-05

CONDITIONS: Dentin Hypersensitivity
Keywords: dentin sensitivity; tooth abrasion; Ca-hydroxyapatite; fluoroapatite; Mg-Zn-hydroxyapatite
MeSH Terms: conditions — Dentin Sensitivity; Tooth Abrasion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - HAP-containing toothpaste (Active Comparator): The use of HAP-containing toothpaste twice daily (using standardised toothbrushing technique) for 4 weeks.
  Toothpaste composition: Aqua, Sorbitol, Hydrated Silica, Glycerin, Hydroxyapatite, Cellulose Gum, Sodium Myristoyl Sarcosinate, Sodium Methyl Cocoyl Taurate, Aroma, Xanthan Gum, Stevia Rebaudiana Extract, Anethole, Tetrasodium Glutamate Diacetate, Tocopheryl Acetate, Eucalyptol, o-Cymen-5-ol, Citric Acid, Vitis Vinifera (Grape) Seed Extract, Tannase, Thymol, Limonene. Fluoride free.
  Interventions: Combination Product: Hygienic procedure (toothbrushing using HAP-containing toothpaste)
- Group 2 - Zn Mg HAP-containing toothpaste (Experimental): The use of Zn Mg HAP-containing toothpaste twice daily (using standardised toothbrushing technique) for 4 weeks.
  Toothpaste composition: Aqua, Sorbitol, Hydrated Silica, Glycerin, Zn-Mg-hydroxyapatite, Cellulose Gum, Sodium Myristoyl Sarcosinate, Sodium Methyl Cocoyl Taurate, Aroma, Xanthan Gum, Stevia Rebaudiana Extract, Anethole, Tetrasodium Glutamate Diacetate, Tocopheryl Acetate, Eucalyptol, o-Cymen-5-ol, Citric Acid, Vitis Vinifera (Grape) Seed Extract, Tannase, Thymol, Limonene. Fluoride free.
  Interventions: Combination Product: Hygienic procedure (toothbrushing using Zn Mg HAP-containing)
- Group 3 - FAP-containing toothpaste (Experimental): The use of FAP-containing toothpaste twice daily (using standardised toothbrushing technique) for 4 weeks.
  Toothpaste composition: Aqua, Sorbitol, Hydrated Silica, Glycerin, Fluorapatite, Cellulose Gum, Sodium Myristoyl Sarcosinate, Sodium Methyl Cocoyl Taurate, Aroma, Xanthan Gum, Stevia Rebaudiana Extract, Anethole, Tetrasodium Glutamate Diacetate, Tocopheryl Acetate, Eucalyptol, o-Cymen-5-ol, Citric Acid, Vitis Vinifera (Grape) Seed Extract, Tannase, Thymol, Limonene.
  Interventions: Combination Product: Hygienic procedure (toothbrushing using FAP-containing toothpaste)

INTERVENTIONS:
Combination Product: Hygienic procedure (toothbrushing using HAP-containing toothpaste) — Toothbrushing using standardised technique and pear-sized amount of HAP-containing toothpaste twice daily for 1 month.
  Arms: Group 1 - HAP-containing toothpaste
Combination Product: Hygienic procedure (toothbrushing using Zn Mg HAP-containing) — Toothbrushing using standardised technique and pear-sized amount of Zn Mg HAP-containing toothpaste twice daily for 1 month.
  Arms: Group 2 - Zn Mg HAP-containing toothpaste
Combination Product: Hygienic procedure (toothbrushing using FAP-containing toothpaste) — Toothbrushing using standardised technique and pear-sized amount of FAP-containing toothpaste twice daily for 1 month.
  Arms: Group 3 - FAP-containing toothpaste

SUMMARY:
This will be a double-blind, randomized, three-arm parallel groups study of the effect of toothpastes containing Ca-hydroxyapatite (HAP), Mg-Zn-hydroxyapatite (Zn-Mg-HAP), or fluoroapatite (FAP).

The aim of the study is to compare the effect of toothpastes containing Ca-hydroxyapatite (HAP), fluoroapatite (FAP), and Mg-Zn-hydroxyapatite (Mg-Zn-HAP) on dentin hypersensitivity associated with dental abrasion.

Materials and methods. Thirty consent patients aged 35-45 with dentin hypersensitivity associated with abrasion will be recruited for the study. The study will have 2 phases: preparatory phase (recruitment of the patients, standardization of their oral hygiene protocols, wash-out period, calibration of the researchers and training) and the main part (double-blind, randomized, parallel groups study of toothpastes effect). Patients will be randomly divided into 3 groups (group 1 - toothpastes with Ca-HAP, group 2 - toothpastes with Zn-Mg-HAP, group 3 - toothpastes with FAP). Clinical examination will be performed at the baseline, after 2 and 4 weeks, and will include patient's interview, oral hygiene level assessment (OHI-S), and dentin sensitivity testing (Shiff's index).

The null hypothesis is that there will be no statistically significant differences in dentin sensitivity level between the study groups.

DETAILED DESCRIPTION:
Background: Dentin hypersensitivity (DH) represents a sharp, short pain arising from exposed dentin in response to various stimuli which cannot be ascribed to any other form of dental defect or pathology. The use of toothpastes containing various HAP-formulations has become one of the most common methods for dentin hypersensitivity management. However, there is a paucity of literature concerning the comparison of the effect of different HAP-formulations.

This will be a double-blind, randomized, three-arm parallel groups study of the effect of toothpastes containing Ca-hydroxyapatite (HAP), Mg-Zn-hydroxyapatite (Zn-Mg-HAP), or fluoroapatite (FAP). The groups will include adults with DH diagnosed clinically.

The aim of the study is to compare the effect of toothpastes containing Ca-hydroxyapatite, fluoroapatite, and Mg-Zn-hydroxyapatite on dentin hypersensitivity in patients with dental abrasion. The sample size was determined according to the trial by Vano et al. (2017), where similar design was used. The power was set at 80%, alfa-level was set as 0.05, the means in the study groups were 2.65±0.68 and 1.72. The allocation ratio was equal to 1. The resultant target sample size comprised 10 participants in each group (7 participants according to sample size calculations plus 30% to account for possible drop-out), 30 patients total.

Subjects who meet all inclusion and exclusion criteria will be randomized on Baseline/Screening Visit in a 1:1:1 ratio to the Group 1, 2, or 3 in accordance with a computer-generated schedule prepared by a third-party person, who will not participate in the study.

The study is estimated to complete enrollment within 1 week from study initiation; however, enrollment will remain open until the study goal is met. The duration of this study for each subject will be a maximum of eight (8) weeks: 4 weeks - preparatory period and 4 weeks - intervention period.

Baseline/Screening Visit

* Review the study with the subject and obtain written informed consent
* Assign the subject a unique screening/enrollment number
* Review and record medical history, and medication history to determine eligibility based on inclusion/exclusion criteria
* Record demographics (age, race, ethnicity, gender)
* Document vitals
* Document all current medications, including medications over-the-counter and herbal medications
* Perform physical examination

  * Administer OHI-S and Shiff test.
  * The allocation concealment will be performed by the use of containers numbered by a "third party" (person, who will not participate in the study). The toothpastes in white bottles without any titles will be placed in the containers. The weight of the pastes and bottles in different groups will be the same. The patient on enrolment will receive a sealed container with a toothpaste. Neither patients nor researchers will be aware of the type of a toothpaste received by each patient (double blinding).

Second visit (2 weeks from the baseline visit) - all groups

* Simplified Oral Hygiene index (OHI-S),
* Schiff test for the assessment of enamel sensitivity,
* Assess for adverse events

Third visit (2 weeks from the second visit) = Final Study Visit - all groups

* Simplified Oral Hygiene index (OHI-S),
* Schiff test for the assessment of enamel sensitivity
* Assess for adverse events

Early Termination visit

* Assess for adverse events
* Assess for complications following treatments
* Document all current medications, including medications over-the-counter and herbal medications

Preparatory phase of the study "Wash-out" period and patient training Most recruited patients with DH are using desensitizing products, and a "wash-out" period will be included before subjects enter the main phase of the study. During this time, the potential study population should not use desensitizing, and their home-care regimen and products will be standardized (provision of identical toothpastes and identical soft toothbrushes). Oral hygiene instructions will be given and the compliance with the recommendations will be controlled with weekly visits to the dental office. The participants will be familiarized with the assessment techniques and trial procedures. Initial sensitivity measurements will be made so that erratic and inconsistent responders can be identified and eliminated.

Qualification and calibration of the observers The clinical examinations will be performed by two dentists who are the members of Therapeutic Dentistry Department, Sechenov University, Moscow, Russia. The examiners will be trained and calibrated to obtain an intra- and inter-examiner agreement of 90%, using Kappa statistics.

The main phase of the study

Thirty people aged 35-45 will be examined and randomly assigned to one of the study groups:

Group 1 will use toothpaste containing HAP. Group 2 will use toothpaste containing Mg-Zn-HAP. Group 3 will use toothpaste containing FAP. The allocation concealment will be performed by the use of containers numbered by a "third party" (person, who will not participate in the study). The toothpastes in white bottles without any titles will be placed in the containers. The weight of the pastes and bottles in different groups will be the same. The patient on enrolment will receive a sealed container with a toothpaste. Neither patients nor researchers will be aware of the type of a toothpaste used.

Treatment protocol The assigned toothpastes and uniform toothbrushes should be used twice daily according to the technique which was used during the preparatory phase of the study.

The patients will use the prescribed toothpastes for a month. Control examinations will be carried out in the following periods: 2 weeks and 4 weeks.

The examination will include:

Simplified Oral Hygiene index (OHI-S), Schiff test for the assessment of enamel sensitivity.

Schiff test is performed to assess enamel sensitivity in all groups as follows: air from air/water syringe is applied perpendicular to the cervical areas of all teeth from a distance of 1 cm for a second. Enamel sensitivity is estimated in accordance with the following criteria:

0 - no reaction,

1. - discomfort but the patient does not insist on stopping the test,
2. - discomfort, accompanied by a request to discontinue the test,
3. - severe pain reaction with pronounced motor reactions aimed at the immediate termination of the test.

Data collection and reporting. Data will be collected at the following points: at baseline, and after 2 and 4 weeks of the assigned toothpastes use.

Data from the study will be maintained for two (2) years after the date the investigation is completed, terminated or until the records are no longer required to support the protocol, whichever date is later. Patient records and data are eligible for inspection and/or copying by applicable regulatory authorities.

Data handling and record keeping Data entry will be completed in the RedCap database (which will cover all the created CRFs). The data will be exported into CSV file format, which will then be used for data analysis. Only de-identified data will be used for data analysis. All hard copy documents will be shredded within five years after completion of the study upon Sponsor approval. Collected de-identified data will be sent to a biostatistician for statistical analysis.

Expected outcomes. It is the expectation that all of the tested toothpastes (HAP, Mg Zn HAP, FAP) will show comparable outcomes. Improvements in tooth hypersensitivity are expected in all groups. Data interpretation and the statistical significance of the results will be described later in this protocol.

Adverse reactions. There is no expectation of any adverse outcomes or reactions due to a patient using the assigned toothpastes. However, hypersensitivity reactions to some of the toothpastes' components are still possible. All participants will be given access to contact info of the investigators. Any adverse reactions should be reported immediately to the investigators.

Reasons for Withdrawal or Termination

The following is a list of possible reasons for study treatment discontinuation:

* Screening Failure
* Subject withdrawal of consent
* Subject is not compliant with study procedures
* Adverse Event that in the opinion of the Investigator would be in the best interest of the subject to discontinue study participation
* Protocol violation requiring discontinuation
* Lost to follow-up All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice.

Statistical analysis plan All analyses will be performed using per-protocol population: the researchers will analyse all subjects who did not substantially deviate from the protocol as to be determined on a per-subject basis by the study principal investigator immediately before database lock.

The normality and sphericity of distribution will be assessed with Shapiro-Wilk and Leven's tests, respectively. The data will be presented as means, standard deviations and 95% confidence intervals for each group at each timepoint of the study. Three-way repeated measures mixed ANOVA model will be performed followed by post-hoc Nemeniy test with adjustment for multiple comparisons. All summary tables will be structured with a column for each timepoint and rows for each toothpaste used in the order (HAP, Zn-Mg-HAP, FAP) and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

ELIGIBILITY:
Inclusion Criteria:

* aged between 35 and 45 years
* signed an approved Informed Consent Form, authorizing the participation in the trial and the use of the results of the trial for educational purposes and for the publication
* the diagnosis of dentin hypersensitivity stated clinically
* a premolar or first molar with an abrasive cervical defect of at least 1 millimeter, and not deeper than 1.5 millimeter, as measured by placing a periodontal probe into the deepest part of the cervical lesion; no mesial, distal or buccal restorations (to avoid confounding hypersensitivity)
* a hypersensitivity score of 2 or higher on the Shiff scale with standardized air-blast stimulation
* no other tooth in the same quadrant exhibiting hypersensitivity

Exclusion Criteria:

* medical and pharmacotherapeutic histories that may compromise the protocol (pregnancy or breastfeeding, allergies to toothpastes ingredients, eating disorders)
* systemic conditions that are etiologic to dentin hypersensitivity (e.g., chronic acid regurgitation)
* excessive dietary or environmental exposure to acids
* periodontal surgery in the preceding 3 months
* orthodontic appliance treatment within previous 3 months
* teeth or supporting structures with any other painful pathology or defects
* teeth restored in the preceding 3 months
* abutment teeth for fixed or removable prostheses
* extensively restored teeth and those with restorations extending into the test area.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-24 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
change in dentin hypersensitivity score according to Shiff's index | 4 weeks after the baseline
  Air from air/water syringe is applied perpendicular to the cervical areas of the tooth from a distance of 1 cm for a second. Enamel sensitivity is estimated in accordance with the following criteria:
  0 - no reaction,
  1. - discomfort but the patient does not insist on stopping the test,
  2. - discomfort, accompanied by a request to discontinue the test,
  3. - severe pain reaction with pronounced motor reactions aimed at the immediate termination of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Polyakova, PhD, Principal Investigator — Sechenov University
Locations (1):
- Institute of Dentistry of Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Makeeva IM, Polyakova MA, Doroshina VY, Turkina AY, Babina KS, Arakelyan MG. [Comparative effectiveness of therapeutic toothpastes with fluoride and hydroxyapatite]. Stomatologiia (Mosk). 2018;97(5):34-40. doi: 10.17116/stomat20189705134. Russian. PMID 30346419
- [Background] Makeeva IM, Budaychieva ZS, Polyakova MA, Margaryan EG, Novozhilova NE, Musiyev AA. [Special aspects of individual oral hygiene in patients with I class gingival recession]. Stomatologiia (Mosk). 2019;98(4):25-28. doi: 10.17116/stomat20199804125. Russian. PMID 31513144
- [Background] Sokhova IA, Doroshina VY, Polyakova MA, Margaryan EG. [Comparative assessment of the effectiveness of toothpastes to reduce hyperesthesia in inflammatory periodontal diseases]. Stomatologiia (Mosk). 2020;99(1):27-32. doi: 10.17116/stomat20209901127. Russian. PMID 32125298
- [Background] Makeeva IM, Polyakova MA, Doroshina VY, Sokhova IA, Arakelyan MG, Makeeva MK. [Efficiency of paste and suspension with nano-hydroxyapatite on the sensitivity of teeth with gingival recession]. Stomatologiia (Mosk). 2018;97(4):23-27. doi: 10.17116/stomat20189704123. Russian. PMID 30199063
- [Background] Polyakova MA, Arakelyan MG, Babina KS, Margaryan EG, Sokhova IA, Doroshina VY, Novozhilova NE. Qualitative and Quantitative Assessment of Remineralizing Effect of Prophylactic Toothpaste Promoting Brushite Formation: A Randomized Clinical Trial. J Int Soc Prev Community Dent. 2020 May 7;10(3):359-367. doi: 10.4103/jispcd.JISPCD_493_19. eCollection 2020 May-Jun. PMID 32802784